CLINICAL TRIAL: NCT00001427
Title: A Phase II Trial of 72-Hour Continuous IV Infusion of 9-Aminocamptothecin With G-CSF Support in Patients With Advanced Ovarian Cancer Previously Treated With Paclitaxel and Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 950056; 95-C-0056
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-01

CONDITIONS: Ovarian Neoplasms
Keywords: Pharmacodynamic Studies; Pharmacokinetics
MeSH Terms: conditions — Ovarian Neoplasms | interventions — 9-aminocamptothecin

INTERVENTIONS:
Drug: 9-aminocamptothecin

SUMMARY:
The objectives of this study are to determine the response rate to 9-AC in patients with advanced ovarian cancer who have recurrent disease after paclitaxel- and cisplatin-based chemotherapy regimens.

DETAILED DESCRIPTION:
This is a Phase II study of 9-aminocamptothecin (9-AC), administered as an intravenous continuous infusion over 72 hours with G-CSF support for patients with advanced refractory ovarian cancer. The objectives of the present study are to determine the response rate to 9-AC in patients with advanced ovarian cancer who have recurrent disease after paclitaxel- and cisplatin-based chemotherapy regimens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Histologically proven, advanced epithelial ovarian cancer.

Histologic confirmation by Pathology Department, NIH, required.

Recurrent disease after paclitaxel and either cisplatin or carboplatin. Combination platinum/paclitaxel acceptable.

Bidimensionally measurable disease on physical exam, radiographs, or peritoneoscopy. Repeat peritoneoscopy after 8 courses of therapy required if documentation of disease was solely by peritoneoscopy.

Laparotomy not required.

No CNS metastasis.

No borderline or mixed histology.

PRIOR/CONCURRENT THERAPY:

See Disease Characteristics.

More than 4 weeks since any prior therapy and recovered.

No prior camptothecin analogue-based chemotherapy.

No prior radiotherapy except intraperitoneal 32-P.

PATIENT CHARACTERISTICS:

Age: 18 and over.

Performance status: ECOG 0-2.

Hematopoietic:

WBC greater than 3,000.

AGC greater than 1,500.

Platelets at least 100,000.

Hemoglobin greater than 9 g/dL OR;

Hematocrit greater than 27 g/dL.

Hepatic:

Bilirubin no greater than 1.5 mg/dL.

Serum transaminases no greater than 2 times normal.

Renal:

24-hour creatinine clearance greater than 45 mL/min (documented by NCI investigator or primary care physician).

Cardiovascular:

No myocardial infarction within 12 months.

No active congestive heart failure.

No heart block.

No arrhythmia requiring medication.

OTHER:

No active uncontrolled infection.

No known HIV positivity.

No second malignancy currently under treatment except: Local basal cell carcinoma of the skin, Cervical carcinoma in situ, Other malignancies (e.g., stage I breast cancer) eligible at the discretion of the principal or associate investigators.

No pregnant women.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1995-01; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Burris HA, Rothenberg ML, Kuhn JG, Von Hoff DD. Clinical trials with the topoisomerase I inhibitors. Semin Oncol. 1992 Dec;19(6):663-9. PMID 1334279
- [Background] Fukuoka M, Niitani H, Suzuki A, Motomiya M, Hasegawa K, Nishiwaki Y, Kuriyama T, Ariyoshi Y, Negoro S, Masuda N, et al. A phase II study of CPT-11, a new derivative of camptothecin, for previously untreated non-small-cell lung cancer. J Clin Oncol. 1992 Jan;10(1):16-20. doi: 10.1200/JCO.1992.10.1.16. PMID 1309380